CLINICAL TRIAL: NCT07287748
Title: A Phase I Trial of the Alpha Particle-emitting Radiopharmaceutical, Af-001, in Patients With Differentiated Thyroid Cancer
Brief Title: A Phase I Trial of Af-001 in Patients With Differentiated Thyroid Cancer
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Alpha Fusion Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: af-001TH; jRCT2031250472 (Other: jRCT)
Record Dates: First submitted 2025-11-20; First posted 2025-12-17 (Actual); Last update posted 2025-12-31 (Actual); Status verified 2025-12

CONDITIONS: DTC - Differentiated Thyroid Cancer
Keywords: DTC; At211; alpha particle-emitting radiopharmaceutical

STUDY DESIGN:
Intervention Model Description: Phase 1a, Phase 1b
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- [211At]NaAt (Experimental): Ph1a: single dose, Ph1b: mutiple dose
  Interventions: Drug: [211At]NaAt

INTERVENTIONS:
Drug: [211At]NaAt — MTD or MTD-1 level to be tested

SUMMARY:
This trial consists of 2 parts, i.e., Part Ia and Ib. The Part Ia is to evaluate the safety and tolerability of a single intravenous dose of af-001 in patients with radically unresectable, recurrent, metastatic differentiated thyroid cancer (papillary carcinoma, follicular carcinoma) refractory to or intolerant of standard-of-care therapy, who have received total thyroidectomy, and to determine the MTD (Maximum tolerated dose).

Part Ib is to evaluate the efficacy and safety of af-001 mutiple doses to patients with radically unresectable, recurrent, metastatic differentiated thyroid cancer (papillary carcinoma, follicular carcinoma), who have received total thyroidectomy and are RAI naïve, randomized into two arms at the determined MTD or the MTD-1 dose level, and to determine the recommended Phase II dose (RP2D)

DETAILED DESCRIPTION:
The Part Ia is a dose escalation part. The Part Ib is a parallel-group comparative study part based on the MTD determined in Part Ia, in which 10 patients each will be randomly assigned to one of two treatment arms, at the MTD for af-001 or the MTD-1 dose level. Patients will be randomly assigned by the enrollment system (allocated at a ratio of 1:1). Random assignment will be performed using the stratified permuted block method. The stratification factor will be the site(s) of metastases.

ELIGIBILITY:
Inclusion Criteria:

<Ia part>

* Patients with differentiated thyroid cancer (papillary carcinoma, follicular carcinoma) after total thyroidectomy.
* Patients with radically unresectable, recurrent, metastatic disease who are judged by the principal investigator or sub-investigator (hereinafter, "principal/sub-investigators") to be refractory to or intolerant of standard-of-care therapy.

<Ib part>

* Patients with radically unresectable, recurrent, metastatic disease who are RAI naive
* Patients with measurable lesions. <Ia/Ib part>
* Patients with an Eastern Cooperative Oncology Group (ECOG) performance status (PS) of 0 to 2 and stable general condition.
* Patients expected to survive for at least 6 additional months based on clinical symptoms and physical examination findings.

Exclusion Criteria:

<Ia/Ib part>

* Patients who need to preserve fertility.
* Females who are pregnant or may be pregnant, breastfeeding patients, or patients or their partners who cannot agree to appropriate contraception.
* Patients with active multiple cancers (synchronous multiple cancers and ectopic double cancers with a disease-free period of <=3 years).
* Patients with uncontrolled active infections.
* Patients who are positive for hepatitis B virus surface (HBs) antigen, hepatitis C virus (HCV) antibodies, or human immunodeficiency virus (HIV) antibodies.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Estimated)
Dates: Start 2026-01-01 (Estimated); Primary Completion 2028-07-31 (Estimated); Study Completion 2028-07-31 (Estimated)

PRIMARY OUTCOMES:
Ph1a: DLT (Dose-limiting toxicity ) based on Japanese translation of the Common Terminology Criteria for Adverse Events (CTCAE) version 5.0, Japan Clinical Oncology Group (JCOG) version | 4 weeks
  DLT evaluation criteria:
  1. Grade ≥4* hematologic toxicity that persists for at least 7 days
  2. Febrile neutropenia regardless of duration
  3. Grade ≥3* thrombocytopenia associated with a bleeding tendency or that requires platelet transfusions
  4. Anemia that requires red blood cell transfusions
  5. Neutropenia associated with infection
  6. Grade ≥3* non-hematologic toxicity that persists for at least 7 days and does not improve with symptomatic treatment, with the following exceptions:
     * Toxicities that can be controlled to Grade ≤2* with maximum supportive herapy
     * Those due to the progression of the primary tumor
  [*: Grades as defined in CTCAE v.5.0 (Japanese translation) JCOG version]
Ph1b: Assessment of tumor reduction effect on MRI or CT scan images | 24 weeks
  Using the "Revised version of the Response Evaluation Criteria in Solid Tumors (RECIST) guidelines version 1.1 (Japanese translation of JCOG version 1.0)" as a reference.

CONTACTS AND LOCATIONS:
Overall Officials: Tahara, Chief, Principal Investigator — National Cancer Center Hospital East
Locations (1):
- National Cancer Center Hospital East, Kashiwa, Japan

IPD SHARING:
Plan to Share IPD: No